CLINICAL TRIAL: NCT06518096
Title: Prediction Model of Microvascular Ischemic Ocular Motor Nerve Palsy and Inflammatory Ocular Motor Nerve Palsy in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: predict-2024
Record Dates: First submitted 2024-07-15; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Neuro-Ophthalmology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to train and validate deep learning systems (DLS) to differentiate between microvascular ischemic ocular motor nerve palsy (v-OMNP) and inflammatory ocular motor nerve palsy (i-OMNP). The method involves using clearly diagnosed v-OMNP and i-OMNP patients from the Department of Neurology database at Beijing Tongren Hospital for further DLS validation, aiding in the differential diagnosis of the aforementioned diseases.

ELIGIBILITY:
The diagnosis of disease is the outcome of the study. The inclusion criteria and exclusion criteria were as follows:

1. Inclusion Criteria:

   * Patients with acute bilateral diplopia within 1 week of onset at admission.

     1. Ischemic Group:
     1. Sudden onset of unilateral CN III, CN IV, or CN VI palsy.
     2. Isolated CN III (without pupil involvement), CN IV, or CN VI palsy.
     3. Presence of vascular risk factors (VRFs).
     4. Significant symptom recovery no earlier than 2 months after onset, with complete (or nearly complete) recovery within 3-6 months.

     2. Inflammatory Group:
     1. Unilateral painful CN III, CN IV, and/or CN VI palsy.
     2. Symptoms (including pain or diplopia signs) significantly improved within 72 hours after treatment with corticosteroids.
     3. MRI of the cavernous sinus showing inflammation, i.e., abnormal widening/enhancement of the affected cavernous sinus with or without granulomatous changes/inflammatory manifestations of adjacent tissues.
2. Exclusion Criteria:

   * 1. Ocular muscle palsy confirmed to be caused by tumors, trauma, infections, stroke, carotid-cavernous fistula, aneurysms, neuromuscular junction disorders, thyroid-related eye diseases, and hereditary diseases at onset or during follow-up.

     2. Presence of other neurological signs in addition to ocular muscle palsy. 3. Severe systemic diseases of the heart, liver, or kidneys, as well as psychiatric and mental illness.

     4. Pregnant or breastfeeding patients. 5. Patients who did not undergo gadolinium-enhanced MRI of the cavernous sinus. 6. Patients younger than 18 years at the time of enrollment. 7. Onset of symptoms more than 1 week before admission. 8. Incomplete data or follow-up period less than 6 months. 9. Disagreements in disease diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cavernous sinus idiopathic inflammation and microvascular ischemic OCN palsy patients admitted to Department of Neurology, Beijing Tongren Hospital, Capital Medical University, between January 2020 and April 2024 were consecutively recruited. In-hospital medical chart records were retrospectively collected. The patients underwent gadolinium-enhanced MRIs of the cavernous sinus. Patients with ophthalmoplegia caused by infections, stroke, tumors, injuries, aplasia, carotid cavernous fistulae, aneurysms, and intracranial hypotension were excluded.
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The diagnosis of acute bilateral diplopia, microvascular ischemic ocular motor nerve palsy or inflammatory ocular motor nerve palsy. | 6 months
  This study aimed to train and validated deep learning systems to differentiate between v-OMNP and i-OMNP. Clinical information, including sex, age at onset, clinical manifestations, inflammatory factors (including C-reactive protein, erythrocyte sedimentation rate, autoimmune antibody in the cerebrospinal fluid), cavernous sinus MRIs, and prognosis, was obtained from hospitalization and follow-up records. The following information was recorded: (1) intracavernous sinus: abnormal side, thickness of cavernous sinus, thickening enhancement, enlargement and enhancement of CN III, CN IV and CN VI, and narrowing of intracavernous internal carotid artery and (2) extracavernous sinus: enhancing adjacent lesions, lacrimal prolapsus, orbital fascial lipocele, eyeball protrusion, thickened eyelids, and dilatation of superior orbital veins.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongren Hospital, Beijing, Beijing Municipality, China